CLINICAL TRIAL: NCT02226562
Title: A Clinical Study Investigating the Efficacy of a Mouthwash in Providing Long Term Relief From Dentinal Hypersensitivity
Brief Title: Clinical Study Investigating the Efficacy of a Mouthwash in Providing Long Term Relief From Dentinal Hypersensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202196; RH02492 (Other: GSK)
Record Dates: First submitted 2014-08-25; First posted 2014-08-27 (Estimated); Results first posted 2015-08-26 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — potassium nitrate; Sodium Fluoride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Potassium nitrate and sodium fluoride (Experimental): 3.0% weight by weight (w/w) potassium nitrate mouthwash with 0.02% sodium fluoride
  Interventions: Drug: Potassium nitrate and sodium fluoride
- Standard fluoride dentifrice (Other): Standard fluoride dentifrice containing 1000 ppm fluoride as sodium monofluorophosphate (SMFP)
  Interventions: Drug: Standard fluoride dentifrice

INTERVENTIONS:
Drug: Potassium nitrate and sodium fluoride — 3.0% w/w potassium nitrate mouthwash with 0.02% sodium fluoride
  Arms: Potassium nitrate and sodium fluoride
Drug: Standard fluoride dentifrice — Standard fluoride dentifrice containing 1000 ppm fluoride as SMFP
  Arms: Standard fluoride dentifrice

SUMMARY:
The aim of this study is to investigate the longitudinal efficacy of a potassium nitrate mouthwash formulation when used as an adjunct to brushing with a standard fluoride dentifrice for the relief of dentinal hypersensitivity (DH) compared to brushing with a standard fluoride dentifrice alone. This will be a single centre, eight week, randomised, examiner blind, two treatment arm, parallel design, stratified (by maximum baseline Schiff Sensitivity Score of the two selected test teeth) study in participants with at least two sensitive teeth that meet all the criteria at the Screening and Baseline visit. Participants will be assessed at Baseline, and at four and eight weeks to monitor clinical efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Participants in good general health, with self-reported history of dentinal hypersensitivity lasting more than 6 months but not more than 10 years.
* Participants with minimum of 20 natural teeth.
* At screening, a minimum of four, non-adjacent teeth.

  1. Teeth showing signs of facial/cervical gingival recession and/or signs of erosion or abrasion.
  2. Teeth with Gingival Index score ≤1 and a clinical mobility of ≤1.
  3. Teeth that are determined to be sensitive by the participant following a 1 second air blast to the cervical margin.

Exclusion Criteria:

* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes.
* Any condition which, in the opinion of the investigator, causes dry mouth.
* Tooth with evidence of current or recent caries, or reported treatment of decay in 12 months of screening.
* In the 8 weeks prior to screening use of an oral care product indicated for the relief of DH.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 191 (Actual)
Dates: Start 2014-09-02; Primary Completion 2014-12-01 (Actual); Study Completion 2014-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fort Wayne, Indiana, United States

REFERENCES:
- [Derived] Hall C, Sufi F, Milleman JL, Milleman KR. Efficacy of a 3% potassium nitrate mouthrinse for the relief of dentinal hypersensitivity: An 8-week randomized controlled study. J Am Dent Assoc. 2019 Mar;150(3):204-212. doi: 10.1016/j.adaj.2018.10.023. PMID 30803493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited at a clinical site in the USA
Groups:
- Dentifrice Plus Oral Rinse: 3.0% weight by weight (w/w) potassium nitrate oral rinse with 0.02% sodium fluoride dentifrice
- Dentifrice Alone: Dentifrice containing 1000 parts per million (ppm) fluoride as sodium monofluorophosphate (SMFP)
Period: Overall Study
Arm/Group | Dentifrice Plus Oral Rinse | Dentifrice Alone
Started | 95 | 96
Completed | 95 | 95 (Lost to follow up)
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dentifrice Plus Oral Rinse | Dentifrice Alone | Total
Number analyzed (Participants) | 95 | 96 | 191
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.7 (8.62) | 39.7 (8.14) | 40.7 (8.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 79 | 160
  Male | 14 | 17 | 31

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Schiff Sensitivity Score at Week 8
Description: The examiner indicated the participant's response to an evaporaitve air stimulus for each tooth using the Schiff Sensitivity Scale scored as follows - 0: Participant does not respond to air stimulation; 1: responds to air stimulus but does not request discontinuation of stimulus; 2: Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score is indicative of an imrpovement in sensitivity.
Time Frame: Baseline to 8 week
Population: The primary population for efficacy assessment was intent-to-treat (ITT) population.The ITT population comprised of participants, who were randomized, received at least one dose of study treatment and provided at least one post-baseline assessment of efficacy.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Dentifrice Plus Oral Rinse | Dentifrice Alone
Number analyzed (Participants) | 95 | 95
Score on scale | -1.47 (0.065) | -0.37 (0.065)
Statistical Analysis 1: Comparison: Dentifrice Plus Oral Rinse vs Dentifrice Alone; Test type: Superiority or Other; p = 0.0001, ANCOVA — The P-value was less than 0.0001; ANCOVA with a factor for treatment and baseline as covariate; Mean Difference (Net) = -1.10, 95% CI 2-sided [-1.28 to -0.92]

2. Secondary Outcome: Mean Change From Baseline in Schiff Sensitivity Score at Week 4
Description: as for outcome 1
Time Frame: Baseline to 4 week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Dentifrice Plus Oral Rinse | Dentifrice Alone
Number analyzed (Participants) | 95 | 95
Scores on scale | -0.94 (0.719) | -0.31 (0.542)

3. Secondary Outcome: Mean Change From Baseline in Tactile Threshold at Week 8
Description: The examiner assessed the response to tactile sensitivity using a Yeaple probe which allowed application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force was reached. The tactile threshold for each tooth was determined by asking the subject whether the sensation caused discomfort. The pressure setting at which the subject gave two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth. At baseline, the maximum force used was 20g; at all subsequent visits, it was 80g.
Time Frame: Baseline to 8 week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Gram(g)
Arm/Group | Dentifrice Plus Oral Rinse | Dentifrice Alone
Number analyzed (Participants) | 95 | 95
Gram(g) | 31.32 (27.869) | 3.74 (13.188)

4. Secondary Outcome: Mean Change From Baseline in Tactile Threshold at Week 4
Description: as for outcome 3
Time Frame: Baseline to 4 week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Gram (g)
Arm/Group | Dentifrice Plus Oral Rinse | Dentifrice Alone
Number analyzed (Participants) | 95 | 95
Gram (g) | 14.11 (21.276) | 0.74 (4.434)

5. Secondary Outcome: Mean Change From Baseline in Visual Rating Scale (VRS) at Week 8
Description: Participants rated the intensity of their response to an evaporative air stimulus using a 10 point VRS scale with 1 indicating 'no pain' and 10 indicating 'Intense pain'. A reduction in the score is indicative of an improvement in sensitivity.
Time Frame: Baseline to 8 week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Dentifrice Plus Oral Rinse | Dentifrice Alone
Number analyzed (Participants) | 95 | 95
Score on scale | -3.05 (2.038) | -1.05 (1.673)

6. Secondary Outcome: Mean Change From Baseline in VRS at Week 4
Description: as for outcome 5
Time Frame: Baseline to 4 week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Dentifrice Plus Oral Rinse | Dentifrice Alone
Number analyzed (Participants) | 95 | 95
Score on scale | -1.64 (1.651) | -0.86 (1.295)

ADVERSE EVENTS:
Time Frame: Upto 8 weeks
Arm/Group | Dentifrice Plus Oral Rinse | Dentifrice Alone
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/96
Other Adverse Events (participants affected / at risk) | 11/95 | 7/96
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dentifrice Plus Oral Rinse (N=95) | Dentifrice Alone (N=96)
Sensitivity of teeth (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Device failure (General disorders) | 0 (0) | 1 (1)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.